CLINICAL TRIAL: NCT01532024
Title: Phase 1 Exploratory Clinical Study of Microdosing NAP for Optical Molecular Imaging in Human Lungs in Healthy Volunteers and in Patients With Acute Lung Injury in Intensive Care
Brief Title: Exploratory Clinical Study of Neutrophil Activation Probe (NAP) for Optical Molecular Imaging in Human Lungs
Acronym: NAP
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Edinburgh (Other)
Collaborators: Medical Research Council (Other Government)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: NAP; 2011-006169-17 (EudraCT Number)
Record Dates: First submitted 2012-01-12; First posted 2012-02-13 (Estimated); Last update posted 2019-11-05 (Actual); Status verified 2019-11

CONDITIONS: Acute Lung Injury
Keywords: Optical Imaging; Neutrophil; Elastase; Molecular Imaging; Acute Lung Injury; ARDS
MeSH Terms: conditions — Acute Lung Injury

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Healthy Volunteers (Experimental): Delivery of intrapulmonary NAP Dose escalation from 5 mcgs to 80mcgs
  Interventions: Other: Microdose of NAP
- Pulmonary Infiltrate in ICU (Experimental): Delivery of NAP (80mcgs) to ventilated patients with pulmonary infiltrates
  Interventions: Other: Microdose of NAP
- Patients with Bronchiectasis (Experimental): Delivery of NAP (80mcgs) to patients with bronchiectasis
  Interventions: Other: Microdose of NAP

INTERVENTIONS:
Other: Microdose of NAP — Delivery of NAP at microdose (<100mcg) by direct pulmonary administration followed by fibreoptic confocal microendoscopy

SUMMARY:
Seriously ill patients may develop a complication called acute lung injury (ALI), a form of inflammation in which lung tissue is filled by fluid containing white blood cells called neutrophils. ALI is common and is often fatal (for example in the USA it is estimated that 190,000 patients develop ALI per annum, of whom 75,000 die). No pharmacological treatment has been shown to improve ALI.

Data from animal models and patients strongly suggest that neutrophils are central to disease progression. However no bedside methods exist to rapidly and accurately determine in seriously ill patients, if neutrophils are present and if they are releasing damaging enzymes such as elastase. As such, the investigating team have developed and synthesised to clinical grade, an imaging agent called NAP (Neutrophil Activation Probe) that detects activated neutrophils and also the damaging enzyme, human neutrophil elastase (HNE). The investigators have extensively tested NAP in animal models for efficacy and safety. It reliably detects activated neutrophils and is not toxic.

NAP is a small molecule that is delivered in tiny doses (called microdoses) to areas of inflammation in human lungs through a bronchoscope. The activity of NAP is visualised by imaging though a tiny camera that is also introduced through the bronchoscope. This camera system is now widely used throughout the world in over 150 sites.

The investigators therefore aim to test the utility and safety of NAP in an exploratory clinical study. The study involves the delivery of NAP to 6 healthy volunteers followed by delivering NAP to 3 patients in ICU with pulmonary infiltrates and 6 patients known to have bronchiectasis.

In the healthy volunteers study, healthy male volunteers recruited from the University of Edinburgh will be invited to participate.

In the ICU study, patients will be recruited from the ICU in the Royal Infirmary of Edinburgh.

In the bronchiectasis study, patients will be recruited from the respiratory service in NHS Lothian.

If the study (which is supported by the Medical Research Council) demonstrates safety and also the ability to image activated neutrophils, the investigators intention is to design future studies in patients with ALI.

DETAILED DESCRIPTION:
Acute lung injury (ALI)/adult respiratory distress syndrome (ARDS) is clinically important (16% of mechanically ventilated patients acquire ALI, of whom one third die), yet no pharmacological therapy has been shown to impact significantly on outcome. This is in part due to inadequate stratification of patients with neutrophil predominant ALI/ARDS and the inability to determine disease activity and hence target therapy.

Molecular Imaging (MI) offers a potential strategy to visualize neutrophil activity in vivo in situ. Indeed FDG PET has been used to image neutrophil activity but it is not a bedside modality, and moving critically ill patients to remote scanners is dangerous and expensive and there there are currently no bedside 'smart' MI solutions that can guide, at the cellular/functional level, the diagnostic or therapeutic pathway in patients with inflammatory lung disease. Indeed, in ICU, there is a specific need to rapidly diagnose patients with deteriorating gas exchange, particularly those with chest X-ray (CXR) shadowing. Such CXR infiltrates result from numerous causes including cardiac failure, fluid overload, secondary pneumonia and ALI/ARDS. All require different treatments but, at present, options to distinguish these conditions are severely limited, resulting in empirical 'blunderbuss' antimicrobial therapy and non-correction of the primary condition. There is now a pressing need to rapidly stratify such patients to inform focused implementation of specific targeted therapies.

Activated neutrophils and their histotoxic products, particularly human neutrophil elastase (HNE), have been specifically implicated in the pathogenesis of ALI/ARDS, and there is considerable clinical interest in new drugs in this area. However, there is currently no way of rapidly determining whether new therapeutic candidates are exerting their predicted effects in situ in the human lung prior to embarking upon major clinical trials. Such a solution would inevitably accelerate the pathway of new drugs to clinical application.

The Proposed Solution: probe-based confocal laser endomicroscopy (pCLE) combined with direct intra-pulmonary instillation of microdoses (pharmacologically-inactive and non-toxic) of a highly specific and sensitive 'smartprobe' (NAP) will detect neutrophil activity and the presence of active HNE in the lungs of ventilated ICU patients.

pCLE itself safely provides high-resolution, real-time images of the human lung at cellular resolution in situ. Alone, however, it provides no functional or molecular information. The investigators have therefore embarked on a discovery programme to synthesise highly sensitive smartprobes, detectable by pCLE and specifically directed against key inflammatory events. This provides a new dimension of clinical application for this cutting-edge technology. NAP, the prototype has now been validated in vitro and in vivo where it is effective at a dose of < 10µg and generates a powerful fluorescent signal in < 30 sec. Our pilot study aims are to apply the combined utility of pCLE and NAP in healthy volunteers and patients with inflammatory lung disease. The study will also provide a prototypic foundation that can be applied to future smartprobes, not only in the lung but in any organ accessible to endoscopy.

The primary end-point will be a proof of concept demonstration that this technique can be used to visualise activated neutrophils over background autofluorescence. Other end points include safety. The investigators shall also assess alveolar (by bronchoscopy) neutrophil activation and elastase activity in patients. Demonstration of activated neutrophils by pCLE in ICU would be expected to lead directly to clinical trials in patients with ALI/ARDS.

ELIGIBILITY:
Inclusion Criteria:

* PART A: healthy male volunteers aged between 18 and 40.
* PART B: Ventilated patients over the age of 18 in on ITU with pulmonary infiltrate
* PART C: Male patients diagnosed with bronchiectasis over the age of 18

Exclusion criteria for part A:

1. Age < 18 or >40 years
2. History of any chronic or ongoing acute illness (with particular reference to asthma, upper respiratory tract infection, lower respiratory tract infection, bronchiectasis, congenital heart disease, ischaemic heart disease, valvular heart disease, diabetes mellitus, chronic renal impairment, urinary tract infection)
3. Any current medication
4. Any history of previous reactions to flourescein or any other anaphylaxis
5. Abnormal physical signs detected at cardiorespiratory examination
6. Temperature >37.3 degrees Celsius
7. Oxygen saturation <95% breathing room air
8. Haemoglobin, white cell count or platelet count outside the normal laboratory reference range
9. Blood sodium, potassium, urea, creatinine, bilirubin, alanine aminotransferase, random glucose or C-reactive protein outside the normal laboratory reference range
10. Forced expiratory volume in one second (FEV1) or forced vital capacity (FVC) <80% predicted
11. FEV1:VC ratio <70%
12. Any significant cardiorespiratory abnormality detected on chest x-ray
13. Peripheral venous access insufficient to support 14 gauge cannulae.
14. General practitioner confirmation of eligibility as a healthy volunteer not received
15. Failure to provide suitable identification (passport/driving licence)
16. Refusal to consent to enter details in 'The Over Volunteering Prevention System' (TOPS) database
17. Positive urine drug screen
18. Participation in any other interventional study or less than three months since their last participation in an interventional study
19. Female

Exclusion Criteria for part B

1. Age <18years
2. Any contraindication for bronchoscopy 22,23
3. Refusal for participation by attending consultant
4. Fi02 >70%
5. PEEP>10cm
6. Recent pneumothorax (whilst on ventilator)
7. Any history of previous reactions to flourescein or any other anaphylaxis
8. Participation in any other interventional study or less than three months since their last participation in an interventional study
9. Female

Exclusion criteria for Part C

1. Age <18years
2. Any contraindication with bronchoscopy
3. Refusal for aprticipation by attending consultant
4. Recent pneumothorax (last 4 weeks)
5. Myocardial infarction within preceding 4 weeks
6. Any history of previous reactions to fluorescein or any other anaphylaxis
7. Participation in any other interventional study or less than three months since their last participation in an interventional study.
8. Female

Ages: 18 Years to 60 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2014-10; Primary Completion 2016-09-02 (Actual); Study Completion 2016-09-02 (Actual)

PRIMARY OUTCOMES:
This is an exploratory clinical study. The primary outcome measure is measurement of fluorescence and imaging parameters determined using pCLE and Cellvizio viewer software. | 15 minutes
  Fluorescent amplification of NAP upon exposure to activated neutrophils in lungs of patients with Acute Lung Injury

SECONDARY OUTCOMES:
Safety in part A and part B and initial proof of concept in ICU to detect neutrophil activation. | Within 24 hours of delivery of NAP
  Absence of any adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Kev Dhaliwal, MD, Study Director — University of Edinburgh; David Newby, MD, Principal Investigator — University of Edinburgh; Chris Haslett, MD, Study Chair — University of Edinburgh; Tim Walsh, MD, Principal Investigator — University of Edinburgh
Locations (3):
- United Kingdom (3):
  - Ward 118, Intensive Care, Royal Infirmary of Edinburgh, Edinburgh, Scotland
  - Wellcome Trust Clinical Research Facility, Edinburgh
  - Royal Infirmary of Edinbrugh, Edinburgh

DOCUMENTS (1):
  • Study Protocol (2015-07-27): https://cdn.clinicaltrials.gov/large-docs/24/NCT01532024/Prot_000.pdf